CLINICAL TRIAL: NCT02462226
Title: The-Optimal-Lymph-Flow ™: An e-Health Approach to Enhancing Management of Chronic Pain and Symptoms Related to Lymphedema Among Women Treated for Breast Cancer
Brief Title: Enhancing Management of Chronic Pain and Symptoms Among Women Treated for Breast Cancer (Lymph-Flow)
Acronym: Lymph-Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-00221
Record Dates: First submitted 2015-05-20; First posted 2015-06-04 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Pain; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Pain; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Precaution (Active Comparator): Patients assigned to Education #1 will receive arm precaution self-care strategies. The webpage also has a section entitled "Arm Precautions," representing current patient education that emphasizes precautionary lifestyle behaviors, such as avoidance of repetitive limb movement, lifting weighted objects, needle punctures, blood draw, and the use of compression garments for air travel in the affected limb. Exercises to promote limb mobility will also provided. Only the patients in the control group will be given access to Arm Precautions section.
  Patients will be given access to the website to learn about the arm precaution program.
  Interventions: Behavioral: Arm Precaution
- The-Optimal-Lymph-Flow (Experimental): The Optimal Lymph-Flow™ is the only evidence-based self-care program designed to effectively help women treated for breast cancer manage daily pain and symptoms related to lymphedema. Grounded in research-driven behavioral strategies, the program is premised on empowering, rather than inhibiting, how breast cancer survivors live their lives. It emphasizes "what to do," rather than "what to avoid." It features a safe, feasible and easily-integrated-into-daily-routine of exercises to promote lymph flow and drainage, as well as guidance to maintain an optimal BMI.
  Patients will be given the access to the website to learn about the The-optimal-Lymph-Flow program
  Interventions: Behavioral: The-Optimal-Lymph-Flow

INTERVENTIONS:
Behavioral: The-Optimal-Lymph-Flow — The-Optimal-Lymph-Flow ™ is a web-based educational and behavioral program focusing on self-care strategies to manage pain and symptoms related to lymphedema. The Optimal Lymph-Flow™ is the only evidence-based self-care program designed to effectively help women treated for breast cancer manage daily pain and symptoms related to lymphedema. Grounded in research-driven behavioral strategies, the program is premised on empowering, rather than inhibiting, how breast cancer survivors live their lives. It emphasizes "what to do," rather than "what to avoid." It features a safe, feasible and easily-integrated-into-daily-routine of exercises to promote lymph flow and drainage, as well as guidance to maintain an optimal BMI.
  Arms: The-Optimal-Lymph-Flow
Behavioral: Arm Precaution — The webpage also has a section entitled "Arm Precautions," representing current patient education that emphasizes precautionary lifestyle behaviors, such as avoidance of repetitive limb movement, lifting weighted objects, needle punctures, blood draw, and the use of compression garments for air travel in the affected limb.
  Arms: Arm Precaution

SUMMARY:
The purpose of this research study is to conduct a randomized clinical trial to evaluate the efficacy of the web-based The-Optimal-Lymph-Flow ™ system for managing chronic pain and symptoms related to lymphedema focusing on primary outcomes of pain reduction, secondary outcomes of symptom relief, limb volume difference by infra-red perometer, body mass index, quality of life related to pain.

Recruitment includes 120 patients who will be randomized according to pain/aching/soreness, and tenderness. Participants in the intervention group will be provided the web-based The-Optimal-Lymph-Flow ™ intervention and encourage to access and learn about the program during the 1-4 weeks of the study. Participants in the control group will receive the web-based arm precaution program. All the participants will have monthly online assessment of pain and symptoms at 4 and 8 weeks post-intervention as well as two in-person research visits, that is, prior to intervention and 12 weeks post-intervention.

DETAILED DESCRIPTION:
Despite current advances in cancer treatment, many breast cancer survivors still face long-term post-operative challenges as a result of suffering from daily pain and other distressing symptoms related to lymphedema, i.e. abnormal accumulation of lymph fluid in the ipsilateral upper limb or body.

The purpose of this research study is to conduct a randomized clinical trial to evaluate the efficacy of the web-based The-Optimal-Lymph-Flow ™ system for managing chronic pain and symptoms related to lymphedema focusing on primary outcomes of pain reduction, secondary outcomes of symptom relief, limb volume difference by infra-red perometer, body mass index, quality of life related to pain.

Recruitment includes 120 patients who will be randomized according to pain/aching/soreness, and tenderness. Participants in the intervention group will be provided the web-based The-Optimal-Lymph-Flow ™ intervention and encourage to access and learn about the program during the 1-4 weeks of the study. Participants in the control group will receive the web-based arm precaution program. All the participants will have monthly online assessment of pain and symptoms at 4 and 8 weeks post-intervention as well as two in-person research visits, that is, prior to intervention and 12 weeks post-intervention. The study length for patients is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been surgically treated for breast cancer more than 3 months; healing usually occurs within 3 months of surgical treatment for cancer
2. Patients who report persistent or intermittent pain, including aching, tenderness, soreness;
3. Patients may or may not report any of symptoms related to lymphedema (i.e. swelling, heaviness, tightness, firmness, numbness, tingling, stiffness, limb fatigue, limb weakness, and impaired limb mobility of shoulder, arm, elbow, wrist, and fingers);
4. Patients may or may not have a history of lymphedema or have been treated for lymphedema.
5. Patients have Internet access to the web-based program at home or willing to access the web-based program using the computer provided by the researchers at the Cancer Center.
6. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who do not report any pain, including aching, tenderness, and soreness;
2. Patients who have known metastatic disease or other bulk disease in the thoracic or cervical regions;
3. Patients who have lymphedema due to cancer recurrence.
4. Patients with documented advanced cardiac or renal disease.

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
The Lymphedema and Breast Cancer Symptom Experience Index (BCLE-SEI | 12 weeks
  The Lymphedema and Breast Cancer Symptom Experience Index (BCLE-SEI) is a valid and reliable self-report tool to assess pain, including aching, soreness, tenderness, as well as symptoms related to lymphedema (i.e. , arm swelling, breast swelling, chest wall swelling, heaviness, firmness, tightness, stiffness, burning, stabbing numbness, tenderness, stiffness, redness, blistering, and tingling (pins and needles. Each symptom can be treated as categorical variable by choosing a "Yes" or "No" to indicate the presence or absence of a given symptom. Each item can also be rated on a Likert-type scale from 0 (no presence of a given symptom) to 4 (greatest severity of a given symptom). Higher scores indicate more severe symptom presence. A response frame of last three months will be used for all participants to ensure the chronicity of symptom presence.

SECONDARY OUTCOMES:
Limb Volume Difference by Infra-red Perometer. | 12 weeks
  Perometry 350S will be performed on each arm as it is held horizontally. The perometer maps a 3-dimensional graph of the affected and non-affected extremities using numerous rectilinear light beams, and interfaces with a computer for data analysis and storage. A 3-dimensional limb image will be generated and limb volume will be calculated. This optoelectronic method has a standard deviation of 8.9 ml (arm), less than 0.5% of Limb Volume with repeated measuring.
The Pain Impact Questionnaire™ (PIQ-6™) | 12 Weeks
  The Pain Impact Questionnaire™ (PIQ-6™), a reliable and valid six question health survey, will be used to measure pain severity and the impact of pain on an individual's functional health and well-being. The PIQ-6 measures the severity of pain and its impact on work and leisure activities, as well as on emotional well-being within a variety of diseases and general populations. High PIQ-6™ T scores indicate greater pain impact/worse health
Body Weight and Body Mass Index [BMI] | 12 Weeks
  An electrical device (InBody 520, Biospace Co., Ltd) will be used to measure the participants' body weight, BMI is calculated using the formula: weight (kg) / height (m2).
Risk Reduction Behavior Checklist | 12 Weeks
  Risk Reduction Behavior Checklist is a structured self-report checklist that will be used to quantitatively and qualitatively assess patients' practice of self-care behaviors at the study endpoint of 12-week after intervention. The checklist include a list of self-care behaviors that promote lymph flow, e.g. muscle-tightening deep breathing, muscle-tightening pumping, shoulder exercises, large muscle exercises, and having nutrition-balance and portion-appropriate diet, as well as compression therapy for lymphedema.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Fu MR, Axelrod D, Guth AA, Scagliola J, Rampertaap K, El-Shammaa N, Qiu JM, McTernan ML, Frye L, Park CS, Yu G, Tilley C, Wang Y. A Web- and Mobile-Based Intervention for Women Treated for Breast Cancer to Manage Chronic Pain and Symptoms Related to Lymphedema: Results of a Randomized Clinical Trial. JMIR Cancer. 2022 Jan 17;8(1):e29485. doi: 10.2196/29485. PMID 35037883
- [Derived] Fu MR, Axelrod D, Guth A, Scagliola J, Rampertaap K, El-Shammaa N, Fletcher J, Zhang Y, Qiu JM, Schnabel F, Hiotis K, Wang Y, D'Eramo Melkus G. A Web- and Mobile-Based Intervention for Women Treated for Breast Cancer to Manage Chronic Pain and Symptoms Related to Lymphedema: Randomized Clinical Trial Rationale and Protocol. JMIR Res Protoc. 2016 Jan 21;5(1):e7. doi: 10.2196/resprot.5104. PMID 26795447